CLINICAL TRIAL: NCT03832647
Title: Multicentric, Parallel, Randomized, Double Blind Study Under Dermatological Control to Evaluate the Anti-acne Efficacy of a Dermo-cosmetic Product (Fla 688977 33) Associated With the Fixed Combination Adapalene 0.1%/ Benzoyl Peroxide 2.5% Treatment Versus This Treatment Associated With a Standard Moisturizer (Hydréane légère, Cosmétique Active International) During a 12-week Application Period in Male and Female Subjects Presenting With Mild to Moderate Acne
Brief Title: Anti-acne Efficacy of a Dermo-cosmetic Product Associated With the Fixed Combination Adapalene 0.1%/ Benzoyl Peroxide 2.5% Treatment Versus This Treatment Associated With a Standard Moisturizer in Male and Female Subjects Presenting With Mild to Moderate Acne
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vichy Laboratoires (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VCA 18-01; 2018-A02481-54 (Other: Agence National de Sécurité du médicament et des produits de santé)
Record Dates: First submitted 2019-01-25; First posted 2019-02-06 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene, Benzoyl Peroxide Drug Combination; Salicylic Acid

STUDY DESIGN:
Intervention Model Description: 100 subjects per arm
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salicylic acid & Epiduo 0.1%-2.5% Topical Gel (Experimental): Salicylic acid: Once-a-day, on the morning, during 12 weeks.
  Epiduo gel: Once-a-day, on the evening (before bedtime) during 12 weeks.
  Interventions: Combination Product: Epiduo; Drug: Salicylic Acid
- Hydréane légère & Epiduo 0.1%-2.5% Topical Gel (Placebo Comparator): Hydréane légère: Once-a-day, on the morning, during 12 weeks.
  Epiduo gel: Once-a-day, on the evening (before bedtime) during 12 weeks.
  Interventions: Combination Product: Epiduo; Other: Hydréane légère

INTERVENTIONS:
Combination Product: Epiduo — 100 per arm Adapalene/ Benzoyl Peroxide
Drug: Salicylic Acid — Salicylic Acid
  Arms: Salicylic acid & Epiduo 0.1%-2.5% Topical Gel
Other: Hydréane légère — moisturizer
  Arms: Hydréane légère & Epiduo 0.1%-2.5% Topical Gel

SUMMARY:
Study to evaluate the anti-acne efficacy of a dermo-cosmetic associated with the fixed combination Adapalene 0.1%/ benzoyl peroxide 2.5% treatment and to demonstrate that the dermo-cosmetic product can improve the local tolerance of the fixed combination Adapalene 0.1%/ benzoyl peroxide 2.5% treatment

Multi centre, Randomised, Double blind, Controlled, Parallel (100 subjects per arm), Intra-subject & inter subject comparisons

ELIGIBILITY:
Inclusion Criteria:

1. Male and/or female subjects aged 16 to 35 years
2. Subjects presenting with mild to moderate acne (stage 2 or stage 3 with at least 12 inflammatory lesions on face according to the Global Acne Evaluation)
3. Female subjects of child-bearing potential who:

   * use the same reliable hormonal contraceptive method (oral contraceptive, implant, intra-uterine device, patch, cervical cap, vaginal ring and injection) for at least 3 months prior to study inclusion and throughout the study or
   * use a reliable non-hormonal contraceptive method (copper intra-uterine device, condoms, diaphragm, cervical cap and spermicide) for at least 1 month prior to study inclusion and throughout the study or
   * have no sexual intercourse and agreeing not to have any throughout the study or
   * are surgically sterile (oophorectomy, hysterectomy or tubal ligation),
4. Subjects and/or all legal representatives (for minor subjects) who have given written informed consent
5. Subjects who are willing to comply with the study requirements
6. Subjects with Social Security (health insurance) coverage (according to the French requirements)

Exclusion Criteria:

1. Subjects with any systemic disorder or face dermatoses other than acne that would in any way confound interpretation of the study results (e.g. atopic dermatitis, eczema, or psoriasis)
2. Subjects with a condition or receiving a medication and/or with a history of medical/surgical events which, in the opinion of the Investigator, could compromise the safety of the subject or affect the outcome of the study
3. Subjects with a history of skin cancer
4. Female subjects who are pregnant (positive urine pregnancy test) or lactating or who are planning to become pregnant during the study
5. Subjects who have started, stopped or changed of hormonal treatment (contraception, thyroid …) in the 3 months prior the study inclusion
6. Subjects with hypersensitivity to the active substances of Epiduo (Adapalene and/or benzoyl peroxide) or to one of its excipients
7. Subjects who are sensitive to peroxides (oxygenated water)
8. Subjects who have received isotretinoin treatment in the 6 months prior to study inclusion
9. Subjects who have been exposed to excessive UV light (natural or artificial) in the 1 month prior to the study inclusion or having planned excessive UV light exposure during the study (e.g. ski holidays, holidays in the tropics…)
10. Subjects who have used systemic drugs for more than 3 consecutive days related to antibiotics, anti-inflammatory, corticoids, anti-acneic in the 4 weeks prior to study inclusion
11. Subjects who have used topical drugs for more than 3 consecutive days related to antibiotics, anti-inflammatory, corticoids, anti-acneic in the 2 weeks prior to study inclusion
12. Subjects who have used scrub, anti-seborrheic topical cosmetic products and/or who have applied self-tanning products on face in the 1 week prior the study inclusion
13. Subjects who have applied cosmetic products for more than 5 consecutive days with alpha hydroxyl-acids, vitamin C, hyaluronic acids in the 1 week prior the study inclusion
14. Subjects having washed the face and/or the hair the day of the study inclusion (only water is accepted the morning of the study inclusion)
15. Subjects having applied any topical products on face (including make-up) the day of the study inclusion
16. Subjects who have planned a major surgery during the study requiring hospitalization under general anesthesia and the use of systemic or topical drugs (e.g. antibiotics, anti-inflammatory) for more than 1 week
17. Subjects who declare to be deprived of their freedom by administrative or legal decision or who are under guardianship
18. Subjects who cannot be contacted by telephone in case of emergency
19. Subjects belonging to the staff of the study centre
20. Subjects in an exclusion period or participating in another biomedical research study

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-17 (Actual)

PRIMARY OUTCOMES:
Evaluation of the anti-acne efficacy 1 (number of the retentional and inflammatory lesions) | Week 0 (baseline) and Week 12 (final time point)
  Change in the number of the retentional (open & closed comedones) and inflammatory lesions (papulae, pustulae & nodules (if applicable)) on face after a 12-week application period At Week 0 (before any application) and Week 12 (after a 12-week application period), a counting of the retentional (open & closed comedones) and inflammatory lesions (papulae, pustulae & nodules (if applicable)) will be performed by a Dermatologist.
  The counting will be broken down on several parts of the face (forehead, left and right cheeks and chin).

SECONDARY OUTCOMES:
Evaluation of the anti-acne efficacy 2 (number of the retentional and inflammatory lesions) | Week 4 and Week 8 (intermediary times point)
  Change in the number of the retentional (open & closed comedones) and inflammatory lesions (papulae, pustulae & nodules (if applicable)) on face after 4 and 8-week application period At Week 4 (after a 4-week application) and Week 8 (after a 8-week application period), a counting of the retentional (open & closed comedones) and inflammatory lesions (papulae, pustulae & nodules (if applicable)) will be performed by a Dermatologist.
  The counting will be broken down on several parts of the face (forehead, left and right cheeks and chin).
Change in the acne stage on face according to the Global Acne Evaluation scale after 4, 8 and 12-week application period | Week 0 (baseline), Week 4 and Week 8 (intermediary times point) and Week 12 (final time point)
  At Week 0 (before any application), Week 4 (after a 4-week application period), Week 8 (after an 8-week application period) and Week 12 (after a 12-week application period), determination of the acne stage will be performed by the Dermatologist according to the Global Acne Evaluation scale (score min:0 to score max:5). More the score decreased, more the treatment is efficient.
Change in the residual marks visibility after 4, 8 and 12-week application period | Week 0 (baseline), Week 4 and Week 8 (intermediary times point) and Week 12 (final time point)
  At Week 0 (before any application), Week 4 (after a 4-week application period), Week 8 (after an 8-week application period) and Week 12 (after a 12-week application period), the residual marks visibility of acne (hyperpigmentation) will be assessed under the same conditions by the Dermatologist using the scale below which include 10 grades (0: absence to 9:numerous). More the score decreased, more the treatment is efficient.
Change in the pores visibility after 4, 8 and 12-week application period | Week 0 (baseline), Week 4 and Week 8 (intermediary times point) and Week 12 (final time point)
  At Week 0 (before any application), Week 4 (after a 4-week application period), Week 8 (after an 8-week application period) and Week 12 (after a 12-week application period), the pores visibility will be assessed under the same conditions by the Dermatologist using the scale below which include 10 grades (0: absence to 9:numerous). More the score decreased, more the treatment is efficient.
Change in the skin shininess after 4, 8 and 12-week application period | Week 0 (baseline), Week 4 and Week 8 (intermediary times point) and Week 12 (final time point)
  At Week 0 (before any application), Week 4 (after a 4-week application period), Week 8 (after an 8-week application period) and Week 12 (after a 12-week application period), the skin shininess will be assessed under the same conditions by the Dermatologist using the scale below which include 10 grades (0: absence to 9:high). More the score decreased, more the treatment is efficient.
Change in skin greasiness after 4, 8 and 12-week application period | Week 0 (baseline), Week 4 and Week 8 (intermediary times point) and Week 12 (final time point)
  At Week 0, Week 4, Week 8 and Week 12, instrumental measurements will be performed by a technician/a nurse.
  The CL measurements (quantity of sebum (casual level)) will be taken using a SEBUMETER®.
  The unit is in µg sebum/cm² of the skin. Only one measurement per subject will be taken in the middle of the forehead. More the value decreased, less the skin is greasy.
Change in skin moisturizing after 4, 8 and 12-week application period | Week 0 (baseline), Week 4 and Week 8 (intermediary times point) and Week 12 (final time point)
  At Week 0, Week 4, Week 8 and Week 12, instrumental measurements will be performed by a technician/a nurse.
  The measurements will be taken using a CM 825 PC CORNEOMETER®. The hydratation values are expressed in arbitrary units ranging from approximately 0 to 120.
  Three measurements per subject will be taken on the right cheekbone. More the value increased, more the skin is moisturize.
Change in skin ph after 4, 8 and 12-week application period | Week 0 (baseline), Week 4 and Week 8 (intermediary times point) and Week 12 (final time point)
  At Week 0, Week 4, Week 8 and Week 12, instrumental measurements will be performed by a technician/a nurse.
  The measurements will be taken using a SKIN PH METER 900®. The result will be expressed in pH units. Only one measurement per subject will be taken on the left cheek, near to the side of the nose. More the value decreased, more the ph is acid.
Total number of hair follicles per cube at a mean depth of 38 µm after a 12-week application period | Week 0 (baseline) and Week 12 (final time point)
  At Week 0 and Week 12, instrumental measurements will be performed by investigator at CHU Nantes.
  Confocal images are obtained by analyzing the reflection of a diode laser in the skin. The lens will be directly applied onto the selected skin area (on 3 nonlesional skin area: forehead, right temple and right mandibular).
  Confocal images will be analyzed by two confocal microscopy experts.
Diameter of the infundibulum in µm after a 12-week application period | Week 0 (baseline) and Week 12 (final time point)
  At Week 0 and Week 12, instrumental measurements will be performed by investigator at CHU Nantes.
  Confocal images are obtained by analyzing the reflection of a diode laser in the skin. The lens will be directly applied onto the selected skin area (on 3 nonlesional skin area: forehead, right temple and right mandibular).
  Confocal images will be analyzed by two confocal microscopy experts.
Aspect of the border (thickness) (number and percentage) after a 12-week application period | Week 0 (baseline) and Week 12 (final time point)
  At Week 0 and Week 12, instrumental measurements will be performed by investigator at CHU Nantes.
  Confocal images are obtained by analyzing the reflection of a diode laser in the skin. The lens will be directly applied onto the selected skin area (on 3 nonlesional skin area: forehead, right temple and right mandibular).
  Confocal images will be analyzed by two confocal microscopy experts.
Onion like appearence (number and percentage) after a 12-week application period | Week 0 (baseline) and Week 12 (final time point)
  At Week 0 and Week 12, instrumental measurements will be performed by investigator at CHU Nantes.
  Confocal images are obtained by analyzing the reflection of a diode laser in the skin. The lens will be directly applied onto the selected skin area (on 3 nonlesional skin area: forehead, right temple and right mandibular).
  Confocal images will be analyzed by two confocal microscopy experts.
Presence of amorphous material into the infundibulum (number and percentage) after a 12-week application period | Week 0 (baseline) and Week 12 (final time point)
  At Week 0 and Week 12, instrumental measurements will be performed by investigator at CHU Nantes.
  Confocal images are obtained by analyzing the reflection of a diode laser in the skin. The lens will be directly applied onto the selected skin area (on 3 nonlesional skin area: forehead, right temple and right mandibular).
  Confocal images will be analyzed by two confocal microscopy experts.
Signs of inflammation (number and percentage) after a 12-week application period | Week 0 (baseline) and Week 12 (final time point)
  At Week 0 and Week 12, instrumental measurements will be performed by investigator at CHU Nantes.
  Confocal images are obtained by analyzing the reflection of a diode laser in the skin. The lens will be directly applied onto the selected skin area (on 3 nonlesional skin area: forehead, right temple and right mandibular).
  Confocal images will be analyzed by two confocal microscopy experts.
Vascularization (number and percentage) after a 12-week application period | Week 0 (baseline) and Week 12 (final time point)
  At Week 0 and Week 12, instrumental measurements will be performed by investigator at CHU Nantes.
  Confocal images are obtained by analyzing the reflection of a diode laser in the skin. The lens will be directly applied onto the selected skin area (on 3 nonlesional skin area: forehead, right temple and right mandibular).
  Confocal images will be analyzed by two confocal microscopy experts.
Presence of Demodex mites (number and percentage) after a 12-week application period | Week 0 (baseline) and Week 12 (final time point)
  At Week 0 and Week 12, instrumental measurements will be performed by investigator at CHU Nantes.
  Confocal images are obtained by analyzing the reflection of a diode laser in the skin. The lens will be directly applied onto the selected skin area (on 3 nonlesional skin area: forehead, right temple and right mandibular).
  Confocal images will be analyzed by two confocal microscopy experts.
Analysis of the efficacy on the skin quality using a questionnaire | Week 12 (final time point)
  Subjects will complete an efficacy questionnaire at the last visit (after a 12-week application period of the Investigational Product (cosmetic product & drug)).
  The following items will be evaluated by the subjects:
  1. Imperfections are less visible
  2. The skin is cleansed/purified
  3. The complexion is homogeneous / uniform
  4. The skin is comfortable
  5. The skin is like hydrated
  6. The skin is smoother
  7. The skin is softer
  8. The skin is suppler
  9. The skin is less brilliant
  10. The skin is matified
  11. Excess sebum is reduced
  12. The skin has a matte touch
  13. The pores of the skin are tightened
  14. Redness of the skin are reduced
  15. The skin texture is refined
  16. The marks of the skin are less visible
  The following scale will be used:
  * Agree ("D'accord")
  * Somewhat agree ("Plutôt d'accord")
  * Neither agree, nor disagree ("Ni d'accord ni pas d'accord")
  * Somewhat disagree ("Plutôt pas d'accord")
  * Disagree ("Pas d'accord")
Analysis of the local tolerance using clinical assessments | Week 0 (baseline), Week 4 and Week 8 (intermediary times point) and Week 12 (final time point)
  At Week 0 (before any application), Week 4 (after a 4-week application period), Week 8 (after an 8-week application period) and Week 12 (after a 12-week application period), a clinical assessment of the face skin condition will be performed by the Dermatologist:
  * Physical signs: erythema, dryness and scaling
  * Functional signs*: tightness, prickling, itching, burning sensation and others
  The following scale will be used:
  Rating 0: none ("absence") Rating 1: slight ("léger") Rating 2: moderate ("modéré") Rating 3: severe ("sévère")
  * During the study, the subjects will have to record any skin discomfort, intensity (slight, moderate or severe) and duration in their daily log. Functional signs will be assessed by the Dermatologist from a review of the daily log and interrogatory of the subject.
  In addition, at W12 (after a 12-week application period), the Dermatologist and the subject.
Products overall tolerance appreciation by the Dermatologist and the subject | Week 12 (final time point)
  In addition, at Week 12 (after a 12-week application period), the Dermatologist and the subject will state about the overall tolerance of the IP (cosmetic product & drug) based on rating scale:
  * Excellent tolerance
  * Good tolerance
  * Medium tolerance
  * Poor tolerance
Analysis of the cosmetic acceptability using a questionnaire | Week 12 (final time point)
  Subjects will complete a cosmetic acceptability questionnaire concerning the cosmetic product at the last visit.
  The following items will be evaluated by the subjects:
  1. The product is easy to spread
  2. The product is easy to apply
  3. The product penetrates quickly
  4. The color of the product is pleasant
  5. The scent of the product is pleasant
  6. The aspect of the product is pleasant
  7. The texture of the product is pleasant
  8. The texture is comfortable
  9. The product doesn't leave the skin sticky
  10. The product doesn't leave a greasy film on the skin
  11. The product leaves a silky effect
  12. The product does not go noodles
  The following scale will be used:
  * Agree ("D'accord")
  * Somewhat agree ("Plutôt d'accord")
  * Neither agree, nor disagree ("Ni d'accord ni pas d'accord")
  * Somewhat disagree ("Plutôt pas d'accord")
  * Disagree ("Pas d'accord")
Evaluation of the skin microbiota using sampling (if applicable) | Week 0 (baseline) and Week 12 (final time point)
  At Week 0 and at Week 12, microbiota sampling will be performed by the same sampler (technician/nurse).
  Skin microbiota sample will be collected on one test site of 4 cm2 on the middle of the left cheek and using aseptic techniques under sterile airflow generated by a portable hood.
  According to the results of the primary variable, the Sponsor will decide to go ahead with the microbiota analysis which will be done by INRA Transfert.
  DNA will be extracted from the swabs. PCR amplification will be performed for each DNA sample. DNA will be PCR amplified. Cleaned pools will be sequenced on the Illumina MiSeq platform.
  Sequences will be then de-replicated and a database containing one sequence for each operational taxonomic unit will be generated.
  Interpretation of these results will be done by Mercurialis.
Analysis of the number of subject with adverse event related to the study product | From Week 0 (baseline) to Week 12 (final time point)
  Adverse Events will be collected during all the study from Week 0 to Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- INTERTEK, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bouloc A, Roo E, Imko-Walczuk B, Moga A, Chadoutaud B, Dreno B. A skincare combined with combination of adapalene and benzoyl peroxide provides a significant adjunctive efficacy and local tolerance benefit in adult women with mild acne. J Eur Acad Dermatol Venereol. 2017 Oct;31(10):1727-1731. doi: 10.1111/jdv.14379. Epub 2017 Jul 7. PMID 28573779
- [Result] Muguet Guenot L, Vourc'h Jourdain M, Saint-Jean M, Corvec S, Gaultier A, Khammari A, Le Moigne M, Boisrobert A, Paugam C, Dreno B. Confocal microscopy in adult women with acne. Int J Dermatol. 2018 Mar;57(3):278-283. doi: 10.1111/ijd.13910. Epub 2018 Jan 25. PMID 29369333
- [Result] Gollnick HP, Bettoli V, Lambert J, Araviiskaia E, Binic I, Dessinioti C, Galadari I, Ganceviciene R, Ilter N, Kaegi M, Kemeny L, Lopez-Estebaranz JL, Massa A, Oprica C, Sinclair W, Szepietowski JC, Dreno B. A consensus-based practical and daily guide for the treatment of acne patients. J Eur Acad Dermatol Venereol. 2016 Sep;30(9):1480-90. doi: 10.1111/jdv.13675. Epub 2016 May 14. PMID 27177989
- [Result] Nast A, Dreno B, Bettoli V, Bukvic Mokos Z, Degitz K, Dressler C, Finlay AY, Haedersdal M, Lambert J, Layton A, Lomholt HB, Lopez-Estebaranz JL, Ochsendorf F, Oprica C, Rosumeck S, Simonart T, Werner RN, Gollnick H. European evidence-based (S3) guideline for the treatment of acne - update 2016 - short version. J Eur Acad Dermatol Venereol. 2016 Aug;30(8):1261-8. doi: 10.1111/jdv.13776. No abstract available. PMID 27514932
- [Result] Zaenglein AL, Pathy AL, Schlosser BJ, Alikhan A, Baldwin HE, Berson DS, Bowe WP, Graber EM, Harper JC, Kang S, Keri JE, Leyden JJ, Reynolds RV, Silverberg NB, Stein Gold LF, Tollefson MM, Weiss JS, Dolan NC, Sagan AA, Stern M, Boyer KM, Bhushan R. Guidelines of care for the management of acne vulgaris. J Am Acad Dermatol. 2016 May;74(5):945-73.e33. doi: 10.1016/j.jaad.2015.12.037. Epub 2016 Feb 17. PMID 26897386

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-07): https://cdn.clinicaltrials.gov/large-docs/47/NCT03832647/Prot_SAP_000.pdf